CLINICAL TRIAL: NCT03781895
Title: Effect of Vitamin D3 on Lung Function and Exercise Tolerance in D3 Deficient COPD Patients
Brief Title: Effect of Vitamin D3 on Lung Function and Exercise Tolerance in COPD Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh (Other)
Responsible Party: Principal Investigator, Samia Hassan, Principal investigator, Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: BSMMU/2016/11228
Record Dates: First submitted 2018-12-11; First posted 2018-12-20 (Actual); Last update posted 2019-01-10 (Actual); Status verified 2019-01

CONDITIONS: Stable COPD Patients
Keywords: COPD; VitaminD3; 6 Minute Walk Distance; Modified BORG scale
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Cholecalciferol; microcrystalline cellulose; Gelatin; stearic acid

STUDY DESIGN:
Intervention Model Description: Two groups of Vitamin D3 deficient stable COPD patients were taken, Group A was given placebo along with standard therapeutic treatment and Group B was given Vitamin D3 along with standard therapeutic treatment
Who Masked: Participant, Care Provider, Investigator
Masking Description: Prospective interventional randomized double blinded study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- A0 (Placebo Comparator): A0- On day 0,before intervention placebo,
  * Microcrystalline Cellulose (303.8gm)
  * Butylated Hydroxy Toluene (0.2mg)
  * Magnesium Stearate (3mg)
  * Gelatin Capsule Shell (1mg)
  weekly,orally,for 90days
  Interventions: Drug: Cholecalciferol
- A90 (Placebo Comparator): A90- On day 90,after intervention placebo,
  * Microcrystalline Cellulose (303.8gm)
  * Butylated Hydroxy Toluene (0.2mg)
  * Magnesium Stearate (3mg)
  * Gelatin Capsule Shell (1mg)
  weekly,orally,for 90days
  Interventions: Drug: Cholecalciferol
- B0 (Active Comparator): B0- On day 0,before intervention cholecalciferol,
  * Cholecalciferol (40,000IU)
  * Microcrystalline Cellulose (58.1 gm)
  * Butylated Hydroxy Toluene ( 0.2mg)
  * Magnesium Stearate (3mg)
  * Gelatin Capsule Shell (1mg)
  80.000IU/week,orally,for 90 days
  Interventions: Drug: Cholecalciferol
- B90 (Active Comparator): B90- On day 90,after intervention cholecalciferol,
  * Cholecalciferol (40,000IU)
  * Microcrystalline Cellulose (58.1 gm)
  * Butylated Hydroxy Toluene ( 0.2mg)
  * Magnesium Stearate (3mg)
  * Gelatin Capsule Shell (1mg)
  80.000IU/week,orally,for 90 days
  Interventions: Drug: Cholecalciferol

INTERVENTIONS:
Drug: Cholecalciferol — • Cholecalciferol (40,000IU),
  ,Microcrystalline Cellulose (58.1 gm), Butylated Hydroxy Toluene ( 0.2mg),Magnesium Stearate (3mg),Gelatin Capsule Shell (1mg)
  Other Names: Microcrystalline Cellulose (58.1 gm); Butylated Hydroxy Toluene ( 0.2mg); Gelatin Capsule Shell (1mg); Magnesium Stearate (3mg)

SUMMARY:
Background: Chronic Obstructive Pulmonary Disease (COPD) is a major cause of morbidity and mortality throughout the world which is a preventable as well as treatable disease. It has some important extra pulmonary effects which may contribute to the magnitude of the severity of this disease. Standard therapeutic treatment alone does not optimize its remedy. Vitamin D3 has been found to improve the physical efficiency of patients with various morbid disorders, including respiratory ailments. Hypothesis:Vitamin D3 administration in stable patients with moderate COPD improves lung function variables along with exercise tolerance.

Objectives: To evaluate the effects of Vitamin D3 on lung functions and exercise tolerance in patients with stable moderate COPD. Methods: For this, a prospective interventional randomized double blinded study will be carried out on 46 vitamin D3 deficient (serum 25 dihidroxycholecalceferol less than 30 ng/ml), male, stable (diagnosed patient, who has not experienced any acute exacerbation , hospitalizations , urgent care visits, or changes in routine medication within 4 weeks prior to study), moderate (post bronchodilator FEV1/FVC<0.70 of predicted value and FEV1=50 to 79% of predicted value) COPD patients (age ≥40 years), who will be selected from the Out Patient Department (OPD) of the National Institute of Diseases of Chest and Hospital (NIDCH) and will be grouped as A (control) and B (study) groups, respectively. All the patients will be again designated as A0, A90 (without D3) and B0, B90 (with D3) for before and after 90 days of follow up. All the participants will be matched in terms of duration of COPD, history of smoking, occupation and socioeconomic status. Along with the standard pharmacological treatment of COPD, the patients of the 'Study group' will be prescribed for 80000 IU of oral vitamin D3 pre week for consecutive 3 months. Along with this, all patients both the groups will be advised to continue ad lib (according to their own choice) diet. At the very 1st day of the study, the lung functions will be assessed by measuring Forced vital capacity (FVC), Forced expiratory volume in one second (FEV1), Forced expiratory ratio (FEV1/FVC%), Peak expiratory flow rate (PEFR) and Forced mid expiratory flow of FVC(FEF25-75%), with a portable digital spirometer. In addition, exercise tolerance will be assessed by change in 6 Minute Walk Distance (6MWD) in 6 Minute Walk Test (6MWT). Changes in peripheral capillary oxygen saturation (SpO2) by Pulse Oximeter and degree of dyspnoea by Modified Borg Scale (MBS) will also be measured both before and after 6MWT to evaluate their change in both the groups. All these variables will be measured again among same 46 patient after 90 days standard pharmacological treatment of COPD with D3 intervention (B group) and also without D3 intervention (A group). For statistical analysis, Chi-square test, independent sample 't' test between two groups, paired Student's 't' test within two specific measurements of different durations of each group ,will be done. In the interpretation of results, ≤0.05 level of probability (p) will be accepted as significant.

DETAILED DESCRIPTION:
1. Introduction:

   Chronic Obstructive Pulmonary Disease (COPD) is one of the major causes of chronic morbidity and mortality throughout the world . Many people suffer from the disease for years and die too early from its complications. COPD is the fourth leading cause of death in adults of United States and also projected to be the third by 2020 .Though it is a preventable and treatable disease, once developed the disease along with its comorbidities cannot be cured. But its progression and morbidity can be reduced.

   The airflow obstruction in this disease is generally persistent as well as progressive .It has two clinical phases (stable phase and exacerbation phase), both of which are associated with inflammation .Independent risk factors for COPD are male gender, advanced age, low socioeconomic status, occupational exposure and cigarette smoking (both active and passive) ,reactivity of airways, occupational factors and air pollution .

   Vitamin D is a steroid important in bone mineralization and calcium homeostasis. The prevalence of vitamin D deﬁciency has been increasing in the general population in recent decades. The majority of circulating 25-hydroxyvitamin D [25(OH)D] is derived from sun exposure with a limited dietary contribution. The increased prevalence of vitamin D deﬁciency is attributed to sun avoidance, indoor lifestyle, use of sunscreen, and decreased intake of vitamin D-containing foods .Because vitamin D is sequestered in adipose tissue, the increasing prevalence of obesity also increases the prevalence of vitamin D deﬁciency .

   Recently, research has found that vitamin D may play a role in multiple chronic diseases such as cancer, autoimmune diseases, infections, and cardiovascular disorders . Vitamin D may also have a role in several diseases involving the respiratory system. Recently some researchers reported that a significant proportion of young COPD patients may have insufficient (20 to 29 ng/ml) serum 25-OHD . Moreover, higher serum vitamin D concentrations, assessed by [25(OH)D], have been associated with better lung function as measured by FEV1 in a large cross-sectional study of the U.S. population . Although the precise connection between vitamin D status and lung function is not clear at this point, it is postulated that vitamin D may improve lung function through its action on regulating inflammation ,inducing antimicrobial peptides , and/or its action on muscles .

   It has also been suggested that, patients with COPD have a high prevalence of vitamin D deficiency, ranging from approximately 30% in mild COPD to over 75% in severe COPD. Particularly for COPD, vitamin D deficiency may enhance chronic airway and systemic inflammation, reduce bacterial clearance, and increase the risk for infectious exacerbations at the same time .

   To provide a quick, acceptable as well as repeatable and reproducible lung function data spirometry is a safe and practical procedure .The ventilatory functions of the lung such as, forced vital capacity (FVC), forced expiratory volume in 1st second (FEV1), FEV1/FVC ratio (FEV1/FVC %), forced mid expiratory flow rate between 25% and 75% of FVC (FEF25-75%) and peak expiratory flow rate (PEFR), can be assessed by spirometry. The indices derived from this forced exhaled maneuver have become the most accurate and reliable way of supporting a diagnosis of COPD . This test should be undertaken in all patients who may have COPD. It is needed to make a confident diagnosis as well as to exclude other diagnoses that may present with similar symptoms. Although spirometry does not fully capture the impact of COPD on a patient's health, it remains the gold standard for diagnosing the disease and monitoring its progression. It is the best standardized most reproducible and most objective measurement of airflow limitation available .

   In addition, oxygen saturation is an indicator of the percentage of hemoglobin saturated with oxygen at the time of the measurement. Peripheral capillary oxygen saturation values obtained from pulse oximetry (SpO2) is one part of a complete assessment of the patient's oxygenation status. Normal oxygen saturation values are 97% to 99% in the healthy individual and of 95% is clinically accepted in a patient with a normal hemoglobin level . This value may vary with the amount of oxygen utilization by the tissues. For example, in some patients, there is a difference in SpO2 values at rest compared with those during activity, such as ambulation or positioning. However it does not reflect the patient's ability to ventilate .

   Moreover, dyspnea is one of the most significant symptoms occurring during the progression of COPD and results from pulmonary hyperinflation, weakness of inspiratory muscles, increased ventilation, voluntary hyperventilation, increased respiratory work load and impaired function of the inspiratory muscles . The evaluation of dyspnea is very important in any chronic respiratory ailment. The effort dyspnea determined at the end of exercise is accepted as the best indicator of dyspnea .There are several scales are available to evaluate dyspnea. Though the interpretation of dyspnea scales depends solely on the statements of the patients, but Modified Borg Scale (MBS) is known to be simple and partially objective, have usually been used to evaluate effort dyspnea in clinical practice .

   Respiratory disease often presents with limited activity level and exercise capacity and reduced exercise tolerance is a hallmark of patients with COPD . In 1963, Balke developed a simple test to evaluate the functional capacity by measuring the distance walked during a period of time. Walk test are typically administered as a means of evaluating functional status, monitoring treatment effectiveness and establishing prognosis. The 6 minutes walk test (6 MWT) is a practical simple test that requires a 30 meter hallway but no exercise equipment or advance training for the observer. The test measures the distance that a person can quickly walk on a flat, hard surface in a period of 6 minutes. The self paced 6 MWT assesses the submaximal level of functional capacity. However, because most activities of daily living are performed at submaximal levels of exertion, the 6 minutes walk distance (6 MWD) may better reflect the functional exercise level for daily physical activities.
2. Rationale:

   Standard therapeutic treatment schedule has a limited role in improving the physical capacity in COPD patients .Various supplementations and extra-therapeutic measures have been tried to improve the functional capacity of the COPD patients . Vitamin D3 supplementation is one of them. The principal goals of adding vitamin D3 in the treatment schedule of these patients are to reduce symptoms and exacerbations, to improve quality of life and to increase physical and emotional participation in everyday activities which may not be adequately addressed by standard pharmacological regime alone for COPD .Recently, a number of studies have shown an association between vitamin D deﬁciency and severity of COPD . In addition in a prospective study, FEV1 was measured in patients with severe and very severe COPD both before and after vitamin D3 supplementation and significant improvement was found .On the other hand, one recent study reported no significant improvement in FVC, FEV1 and FEV1/FVC% in Vitamin D3 insufficient COPD patients after vitamin D3 administration as compared to that of the control group .

   However the volume of information regarding the effect of vitamin D3 administration in COPD patients is not enough for reaching any final conclusion. Moreover, with the best of our knowledge no study have been conducted to observe the effects of this fat soluble vitamin on the spirometric lung function status, oxygen saturation and exercise tolerance in vitamin D3 insufficient, stable patients with moderate COPD.

   Therefore, on the basis of this background the present study has been designed to evaluate the effects of Vitamin D3 on the spirometric lung function status, peripheral capillary oxygen saturation and exercise tolerance in D3 insuffucient, male patients with stable moderate COPD. This study will draw attention of the physicians about the beneficial effects of the vitamin D3 on both pulmonary and extrapulmonary complications in COPD patients.

   Research Question:

   Does vitamin D3 has any effect on lung function and exercise tolerance in stable COPD patients?

   Hypothesis:

   Vitamin D3 administration in stable patients with moderate COPD improves lung function variables along with exercise tolerance.

   Objectives:

   General Objective To evaluate the effects of vitamin D3 administration on lung functions and exercise tolerance in vitamin D3 insufficient male patients with stable moderate COPD.

   Specific Objectives
   * To measure the FVC, FEV1, FEV1/FVC%, PEFR and FEF25-75% of vitamin D3 insufficient male patients with stable moderate COPD, in order to assess their lung function status.
   * To measure the SpO2 at rest, in order to assess the basal oxygenation status in this group of patients.
   * To determine level of dyspnea at rest, in order to assess the basal breathlessness level in the same group of patients
   * To measure the 6MWD of all the patients, in order to assess their functional exercise capacity.
   * To measure both the SpO2 and level of dyspnea again after 6MWT, for the assessment of their exercise tolerance.
   * To measure all these variables after 90 days standard pharmacological treatment with vitamin D3 and also without vitamin D3 in stable COPD patients.
   * To compare the results of baseline and endline.

   Methodology:

   TYPE OF STUDY : Prospective interventional randomized double blinded study PLACE OF STUDY : Department of Physiology, Bangabandhu Sheikh Mujib Medical University (BSMMU), Shahbagh, Dhaka STUDY PERIOD : March 2017 to February 2018 STUDY POPULATION : Stable, moderate COPD patients with vitamin D3 insufficiency.

   SAMPLE SIZE : 46 SAMPLING : Simple random sampling . According to the selection criteria total 46 COPD patients suitable for the aims and objectives of the study, will be enrolled. 46 patients of COPD will be selected by clinician in OPD.

   GROUPING OF THE SUBJECTS :

   Group A (Control group) : 23 D3 insufficient COPD patients without D3 administration A0 : On day 0 A90 : On day 90 Group B (Study group) : 43 (forty three) D3 insufficient COPD patients with D3 administration B0 : On day 0 B90 : On day 90

   Sample size calculation:

   Using the following statistical formula n = (Zα+Zβ) 2 X (σ12+σ22) (μ1-μ2)2

   Here, Using the following statistical formula n = [(Zα+Zβ)2 X (σ12+σ22)] / (μ1-μ2)2 Mean of control, μ1 = 47.1 Mean of study group, μ2 = 67.4 SD of control, σ1 = 26.9 SD of study group, σ2 = 27.5 (Martineau et al. 2015) Type I Error, Zα = 1.96 Type II Error, Zβ = 1.64 (Kirkwood and Sterne 2003) (Kirkwood and Sterne 2003)

   Therefore, n = [(Zα+Zβ)2 X (σ12+σ22)] / (μ1-μ2)2
   * [(1.96+1.64)2 X (26.92 +27.52) / (47.1-67.4)2
   * [12.96 X (756.25+723.61)] / (20.3) 2 = 19178.98 / 412.09 = 46.54 = 47

   Subject Selection:

   After selection of subject the researcher will sit for an interview with the subject. The researcher will at first introduce himself mentioning his institutional affiliation, conflict of interest and will supply address, contact telephone number and information about sponsorship. After that the subject will be thoroughly informed about the objectives and outcome of the study. Brief explanation of the procedure will be given to them. The subject will also be assured if any problem arises during the test; it will be taken care of. The result of the test will be sent to him free of charge and if any abnormality is detected, then appropriate management will be given to him, if possible or will be referred to specific treatment facility as appropriate. He will be encouraged for voluntary participation in a cordial and friendly attitude and will be allowed freedom to withdraw from the study whenever he likes even after participation. They will be informed about the method of confidentiality of their identification. Their identity will be recorded only in questionnaire which will be kept in safe custody with the researcher. It will not enter in the computer and will not go in any publication. No personal identification will be used in data analysis, report writing or publication. They will also be assured that interview time will minimum for maintaining their comfort, some questions will be asked about the personal, family and medical history without any private enquiry. The conflict of interest will be told to him if there is any. After he has understood these entire procedure, if he agrees to participate, then a willingly given informed written consent will be taken from him.

   There is no possibility of any physical, social or mental risk of the respondent. A pretested questionnaire will be filled up by the research assistant.

   All gathered information will be kept secret and only will be used for medical research and analysis.

   SITE OF SAMPLE COLLECTION:

   All the patients will be collected from the Out Patient Department (OPD) of National Institute of Diseases of Chest and Hospital

   STUDY PROCEDURE:

   On the first day of enrollment, the objectives, nature, purpose and potential risk of all the procedures used for the study will be explained in detail to each subject, with a cordial attitude giving emphasis on the benefits he might obtain from this study. He will be encouraged for voluntary participation and will be allowed to withdraw himself from the study even after participation, whenever he felt uneasy. If he agreed to be enrolled in the study, an informed written consent will be taken in a prescribed form . Detailed family history, medical history and thorough physical examination of each patient will be done and all the information will be recorded in a standard data sheet . Then all the patients will be requested to attend the Department of Physiology at 9 am (about 1 and 1/2 hours after his breakfast) on the day of biochemical and spirometric examination.

   On the examination day, 5 ml of venous blood will be collected and taken to the Hematology laboratory as soon as possible for the estimation of serum 25-hydroxycholecalceferol, serum glucose 2 hours after breakfast and serum creatinine. After that his height and weight will be measured and the spirometric lung function test will be done by using a portable spirometer. After getting all the biochemical and spirometric reports the final selection will be done, according to the inclusion and exclusion criteria.

   Subsequently, all the eligible patients will be randomly assigned to either 'Control' or 'Study' groups and will be thoroughly informed about the objectives and detailed study procedure, once again. Then the patients will be examined for the baseline value of all the study variables in Day 1.

   Again after 90 days the study variables will be collected from same 86 patients.

   Vitamin D3

   Ingredient
   * Cholecalciferol (40,000IU)
   * Microcrystalline Cellulose (58.1 gm)
   * Butylated Hydroxy Toluene ( 0.2mg)
   * Magnesium Stearate (3mg)
   * Gelatin Capsule Shell (1mg)

   Dose : 80,000 IU/wk

   Route : Oral

   Placebo : Courtesy of Beximco Pharmaceuticals Limited
   * Bangladesh Ingredient : • Microcrystalline Cellulose (303.8gm)

     * Butylated Hydroxy Toluene (0.2mg)
     * Magnesium Stearate (3mg)
     * Gelatin Capsule Shell (1mg)

   STUDY VARIABLES:

<!-- -->

1. Spirometric variables

   • FVC (L) : Forced Vital Capacity

   • FEV1 (L) : Forced Expiratory Volume in 1st second
   * FEV1/FVC Ratio (%) : Forced Expiratory Ratio
   * PEFR (L/min) : Peak Expiratory Flow Rate
   * FEF 25-75 (L/S) : Forced Expiratory Flow in the middle of FVC
2. Oxygenation variables

   • Resting SpO2 (%) : Resting Peripheral Capillary Oxygen saturation
3. Exercise tolerance variables • 6MWD (meter) : Six Minute Walk Distance • Level of Dyspnea : Modified Borg Scale
4. Hematological variables • 25(OH)D (ng/ml) : 25-hydroxycholecalceferol • PTH (pmol/l) : Parathyroid hormone • Ca2+ (mg/ml) : Ionic calcium • PO43- (mg/ml)

   * Ionic phosphate

     * AP (U/L) : Alkaline Phosphatase

Subsequently a standard therapeutic treatment will be prescribed to all the selected stable moderate COPD patients. In addition, the patients of the 'Study group' will be prescribed for 80000 IU of oral vitamin D3 per week for consecutive 90 days . Along with this, all the patients of both the groups will be advised to continue ad lib (according to their own choice) diet.

Proper education will be given about drug , method of taking medication and medication plan.Afterwards,a good rapport will be built up to take time to time follow up over telephone and visiting patient's place .Schedule appointment ,hotline and follow up will be maintained properly. They will be requested to attend the Department of Physiology again on the 90th day, to have the assessment of all the above-mentioned study variables Any patient, who failed to follow the study procedure exactly during study period, will be dropped and a new one will be included to fulfill the desired total sample number.Thats why extended sample should be taken to fulfill the total sample number.

ELIGIBILITY:
Inclusion Criteria:

* Socioeconomic status: Middle class
* Smoker
* Stable patients of COPD with >1year duration
* Vitamin D3 deficient :

Serum 25-hydroxycholecalciferol, [25(OH)D] level <30ng/ml (Vitamin D Council 2017)

Exclusion Criteria:

* With acute exacerbation of any pulmonary diseases, as,

with acute exacerbation of any cardiac disease, like -

* Uncontrolled systemic hypertension
* Chronic liver disease
* Malignancy
* Use of drugs known to affect vitamin D metabolism within 1 month prior to With biochemical evidence of -
* uncontrolled diabetes mellitus and
* renal insufficiency

All the criteria mentioned above were scrutinized by taking history and clinical examination, except vitamin D3 deficiency, uncontrolled diabetes mellitus and renal insufficiency, which were diagnosed biochemically.

Ages: 40 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2018-02-01 (Actual); Study Completion 2018-02-01 (Actual)

PRIMARY OUTCOMES:
Lung function (Spirometric variables) Forced Vital Capacity(FVC) will be changed | After 90 days FVC will be measured again
  Forced Vital Capacity It is the volume of air that can be expired as forcefully and rapidly as possible after maximal inspiration. In adult male it is about 4.6 liters. The FVC is commonly reduced in obstructive processes such as COPD.Increment of Forced Vital Capacity means improvement in outcome.
Lung function [ Lung function (Spirometric variables): Forced Expiratory Volume in 1st second(FEV1) will be changed | After 90 days FEV1 will be measured again
  Forced Expiratory Volume in 1st second When a person inspires maximally and exhales forcefully, then the volume, which is exhaled in 1st second is known as 'Forced Expiratory volume in 1st second'. It is normally 80% of forced vital capacity .
  Significance- This measurement is much more sensitive index of severity of the obstructive disease .In COPD ,FEV1 is reduced ,Increment of FEV1 indicates improvent in outcome
Lung function (Spirometric variables) Forced Expiratory Ratio [FEV1/FVC Ratio (%)] will be changed | After 90 days FEV1/FVC Ratio will be measured again
  Forced Expiratory Ratio It is the ratio of FEV1 to FVC expressed in percentage. FEV1/FVC ratio = FEV1/FVC×100. It is about 70% or higher.
  Forced Expiratory Ratio is less than 70% in COPD patients.Increment of Forced Expiratory Ratio indicates improvement in outcome
Lung function (Spirometric variables) Peak Expiratory Flow Rate [PEFR (L/min)] will be changed | After 90 days PEFR will be measured again
  Peak Expiratory Flow Rate It is the maximum expiratory rate, beyond which the flow cannot be increased even with greatly increased additional force.
  In adult it is about 400-700 Liter/second.
Lung function (Spirometric variables) Forced Expiratory Flow in the middle of FVC [FEF 25-75 (Liter/Second) ] will be changed | After 90 days FEF 25-75 will be measured again
  Forced Expiratory Flow in the middle of FVC Forced expiratory flow during the middle half of the FVC. Formerly it was called the maximal mid-expiratory flow (MMEF), expressed in liters/second Normal range in male : 1.5-4.5 Liter/second.Increment of Forced Expiratory Flow in the middle of FVC means improvement in outcome.
Lung function (Spirometric variables) Maximum expiratory Flow rate at 25%of the FVC (MEF 75) will be changed | After 90 days MEF 75 will be measured again
  Maximum expiratory Flow rate at 25%of the FVC (MEF 75) Maximum expiratory flow rate when 25% of the FVC remains in the lung to be exhaled and is equivalent to the FEF75 where 75% of the FVC has been exhaled. Expressed in liters/second.
  This is reduced in COPD. Increment in maximum expiratory flow at 25%of the FVC means improvement in outcome
Lung function (Spirometric variables) Maximum expiratory Flow at 50%of the FVC(MEF50) will be changed | After 90 days MEF 50 will be measured again
  Maximum expiratory Flow at 50%of the FVC(MEF50) Maximum expiratory flow rate when 50 % of the FVC remains in the lung to be exhaled and is equivalent to the FEF50 where 50% of the FVC has been exhaled. Expressed in liters/second. This is reduced in COPD.
  Increment in maximum expiratory flow at 50%of the FVC means improvement in outcome.
Lung function (Spirometric variables) Maximum expiratory Flow at 75%of the FVC (MEF25)]will be changed | After 90 days MEF25 will be measured again
  Maximum expiratory Flow at 75%of the FVC (MEF25) Maximum expiratory flow rate when 75% of the FVC remains in the lung to be exhaled and is equivalent to the FEF25 where 25% of the FVC has been exhaled. Expressed in liters/second.This is reduced in COPD.Increment in maximum expiratory flow at 75%of the FVC means improvement in outcome
Exercise Tolerance [Oxygenation variables] Peripheral Capillary Oxygen saturation[SpO2 (%) ] will be changed | After 90 days SpO2 will be measured
  Oxygenation variables Peripheral Capillary Oxygen saturation between 96% to 99% is normal.Peripheral Capillary Oxygen saturation between 96% to 99% means improved outcome
Exercise Tolerance Exercise tolerance variables •Six Minute Walk Distance[6MWD (meter) ]will be changed | After 90 days 6MWD will be measured
  Exercise tolerance variables • Six Minute Walk Distance [6MWD (meter) ] minimum 350m in 6minute at a time(without taking any rest) is standard.The more the distance,the more the better outcome.
Exercise Tolerance variables • Level of Dyspnea : Modified Borg Scale will be changed | After 90 days level of Dyspnea will be measured
  Level of Dyspnea : Modified Borg Scale If the dyspnea score decreases,it means better outcome If the dyspnea score increases,it means outcome is worse
Exercise Tolerance variables Level of fatigue: Modified Borg Scale will be changed | After 90 days level of fatigue will be measured
  Level of fatigue: Modified Borg Scale If the fatigue score decreases,it means better outcome, If the fatigue score increases,it means outcome is worse

CONTACTS AND LOCATIONS:
Overall Officials: Samia Hassan, Principal Investigator — Bangabandhu Sheikh Mujib Medical University and National Institute of Disease of the Chest and Hospital
Locations (1):
- Samia Hassan, Dhaka, Bangladesh

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Agusti AG. COPD, a multicomponent disease: implications for management. Respir Med. 2005 Jun;99(6):670-82. doi: 10.1016/j.rmed.2004.11.006. Epub 2005 Jan 8. PMID 15878483
- [Background] Al Zaabi A, Asad F, Abdou J, Al Musaabi H, Al Saiari MB, Buhussien AS, Nagelkerke N, Soriano JB. Prevalence of COPD in Abu Dhabi, United Arab Emirates. Respir Med. 2011 Apr;105(4):566-70. doi: 10.1016/j.rmed.2010.12.008. Epub 2011 Jan 7. PMID 21216136
- [Background] Atsou K, Chouaid C, Hejblum G. Variability of the chronic obstructive pulmonary disease key epidemiological data in Europe: systematic review. BMC Med. 2011 Jan 18;9:7. doi: 10.1186/1741-7015-9-7. PMID 21244657
- [Background] Afonso AS, Verhamme KM, Sturkenboom MC, Brusselle GG. COPD in the general population: prevalence, incidence and survival. Respir Med. 2011 Dec;105(12):1872-84. doi: 10.1016/j.rmed.2011.06.012. Epub 2011 Aug 17. PMID 21852081
- [Background] Barbu C, Iordache M, Man MG. Inflammation in COPD: pathogenesis, local and systemic effects. Rom J Morphol Embryol. 2011;52(1):21-7. PMID 21424028
- [Background] Biswas S, Hwang JW, Kirkham PA, Rahman I. Pharmacological and dietary antioxidant therapies for chronic obstructive pulmonary disease. Curr Med Chem. 2013;20(12):1496-530. doi: 10.2174/0929867311320120004. PMID 22963552
- [Background] Black PN, Scragg R. Relationship between serum 25-hydroxyvitamin d and pulmonary function in the third national health and nutrition examination survey. Chest. 2005 Dec;128(6):3792-8. doi: 10.1378/chest.128.6.3792. PMID 16354847
- [Background] van de Bool C, Steiner MC, Schols AM. Nutritional targets to enhance exercise performance in chronic obstructive pulmonary disease. Curr Opin Clin Nutr Metab Care. 2012 Nov;15(6):553-60. doi: 10.1097/MCO.0b013e328358bdeb. PMID 23075934
- [Background] Caballero A, Torres-Duque CA, Jaramillo C, Bolivar F, Sanabria F, Osorio P, Orduz C, Guevara DP, Maldonado D. Prevalence of COPD in five Colombian cities situated at low, medium, and high altitude (PREPOCOL study). Chest. 2008 Feb;133(2):343-9. doi: 10.1378/chest.07-1361. Epub 2007 Oct 20. PMID 17951621
- [Background] Dawson-Hughes B, Heaney RP, Holick MF, Lips P, Meunier PJ, Vieth R. Estimates of optimal vitamin D status. Osteoporos Int. 2005 Jul;16(7):713-6. doi: 10.1007/s00198-005-1867-7. Epub 2005 Mar 18. PMID 15776217
- [Background] De Smet K, Contreras R. Human antimicrobial peptides: defensins, cathelicidins and histatins. Biotechnol Lett. 2005 Sep;27(18):1337-47. doi: 10.1007/s10529-005-0936-5. PMID 16215847
- [Background] Eickhoff P, Valipour A, Kiss D, Schreder M, Cekici L, Geyer K, Kohansal R, Burghuber OC. Determinants of systemic vascular function in patients with stable chronic obstructive pulmonary disease. Am J Respir Crit Care Med. 2008 Dec 15;178(12):1211-8. doi: 10.1164/rccm.200709-1412OC. Epub 2008 Oct 3. PMID 18836149
- [Background] Fabricius P, Lokke A, Marott JL, Vestbo J, Lange P. Prevalence of COPD in Copenhagen. Respir Med. 2011 Mar;105(3):410-7. doi: 10.1016/j.rmed.2010.09.019. Epub 2010 Oct 16. PMID 20952174
- [Background] Finkelstein J, Cha E, Scharf SM. Chronic obstructive pulmonary disease as an independent risk factor for cardiovascular morbidity. Int J Chron Obstruct Pulmon Dis. 2009;4:337-49. doi: 10.2147/copd.s6400. Epub 2009 Sep 24. PMID 19802349
- [Background] Forli L, Bjortuft O, Boe J. Vitamin D status in relation to nutritional depletion and muscle function in patients with advanced pulmonary disease. Exp Lung Res. 2009 Aug;35(6):524-38. doi: 10.1080/01902140902763193. PMID 19842836
- [Background] Holick MF, Chen TC. Vitamin D deficiency: a worldwide problem with health consequences. Am J Clin Nutr. 2008 Apr;87(4):1080S-6S. doi: 10.1093/ajcn/87.4.1080S. PMID 18400738
- [Background] Hopkinson NS, Li KW, Kehoe A, Humphries SE, Roughton M, Moxham J, Montgomery H, Polkey MI. Vitamin D receptor genotypes influence quadriceps strength in chronic obstructive pulmonary disease. Am J Clin Nutr. 2008 Feb;87(2):385-90. doi: 10.1093/ajcn/87.2.385. PMID 18258629
- [Background] Ismail M, Hossain MF, Tanu AR, Shekhar HU. Effect of spirulina intervention on oxidative stress, antioxidant status, and lipid profile in chronic obstructive pulmonary disease patients. Biomed Res Int. 2015;2015:486120. doi: 10.1155/2015/486120. Epub 2015 Jan 22. PMID 25685791
- [Background] Jabbari A, Tabasi S, Masrour J. Vitamin D serum level and chronic obstructive lung disease. Caspian J Intern Med. 2013 Winter;4(1):624-6. No abstract available. PMID 24009949
- [Background] Janssens W, Lehouck A, Carremans C, Bouillon R, Mathieu C, Decramer M. Vitamin D beyond bones in chronic obstructive pulmonary disease: time to act. Am J Respir Crit Care Med. 2009 Apr 15;179(8):630-6. doi: 10.1164/rccm.200810-1576PP. Epub 2009 Jan 22. PMID 19164701
- [Background] JACKSON GG, DOWLING HF, SPIESMAN IG, BOAND AV. Transmission of the common cold to volunteers under controlled conditions. I. The common cold as a clinical entity. AMA Arch Intern Med. 1958 Feb;101(2):267-78. doi: 10.1001/archinte.1958.00260140099015. No abstract available. PMID 13497324
- [Background] James PA, Oparil S, Carter BL, Cushman WC, Dennison-Himmelfarb C, Handler J, Lackland DT, LeFevre ML, MacKenzie TD, Ogedegbe O, Smith SC Jr, Svetkey LP, Taler SJ, Townsend RR, Wright JT Jr, Narva AS, Ortiz E. 2014 evidence-based guideline for the management of high blood pressure in adults: report from the panel members appointed to the Eighth Joint National Committee (JNC 8). JAMA. 2014 Feb 5;311(5):507-20. doi: 10.1001/jama.2013.284427. PMID 24352797
- [Background] Kunisaki KM, Niewoehner DE, Singh RJ, Connett JE. Vitamin D status and longitudinal lung function decline in the Lung Health Study. Eur Respir J. 2011 Feb;37(2):238-43. doi: 10.1183/09031936.00146509. Epub 2010 Jul 1. PMID 20595151
- [Background] Kendrick KR, Baxi SC, Smith RM. Usefulness of the modified 0-10 Borg scale in assessing the degree of dyspnea in patients with COPD and asthma. J Emerg Nurs. 2000 Jun;26(3):216-22. doi: 10.1016/s0099-1767(00)90093-x. PMID 10839848
- [Derived] Williamson A, Martineau AR, Jolliffe D, Sheikh A, Janssens W, Sluyter J, Rafiq R, de Jongh R, Griffiths CJ. Vitamin D for the management of chronic obstructive pulmonary disease. Cochrane Database Syst Rev. 2024 Sep 27;9(9):CD013284. doi: 10.1002/14651858.CD013284.pub2. PMID 39329240

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-12-23): https://cdn.clinicaltrials.gov/large-docs/95/NCT03781895/Prot_SAP_000.pdf
  • Informed Consent Form (2019-01-01): https://cdn.clinicaltrials.gov/large-docs/95/NCT03781895/ICF_001.pdf